CLINICAL TRIAL: NCT04532814
Title: Exercise-stimulated Muscle Glucose Uptake in Upper Body Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael D. Jensen, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-002949; R01DK045343 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Upper Body Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study is aimed to determine whether obesity effects muscle glucose utilization during exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean (Other): Control
  Interventions: Other: Exercise
- Obese (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Cycling 60% VO2 max

SUMMARY:
The purpose of this study is to provide the first integrated examination of the interaction between muscle insulin action and exercise-stimulated muscle glucose uptake in obesity from the whole body to the cellular/molecular level.

ELIGIBILITY:
Inclusion Criteria:

For the exercise studies of leg glucose uptake - "insulin sensitive" group:

* Sedentary, normal weight, premenopausal women.
* Sedentary, age-matched normal weight men.
* Weight stable for two (2) months prior to study.
* Willing to provide written, informed consent.
* For the exercise studies of leg glucose uptake - "insulin resistant" group:

For the exercise studies of leg glucose uptake - "insulin resistant" group:

* Upper body obese (UBO) premenopausal women.
* Age-matched upper body obese (UBO) men.
* Weight stable for two (2) months prior to study.
* Willing to provide written, informed consent.

Exclusion Criteria:

* Age < 18 or > 55 years (premenopausal women and age-matched men).
* Use of glucose-lowering agents.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle glucose uptake | 1 hour
  Is exercise induced skeletal muscle glucose uptake different in obese compared to lean adults

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT04532814/ICF_000.pdf